CLINICAL TRIAL: NCT06615947
Title: Clinical Trial to Compare Conventional Multidisciplinary Gait Rehabilitation With the Atalante Self-balancing Walking System in Patients With Multiple Sclerosis
Brief Title: Conventional Multidisciplinary Gait Rehabilitation VR Robotic Self-balancing Based Gait Rehabilitation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Multiple Sclerosis Center of Catalonia (Other)
Responsible Party: Principal Investigator, Edwin Roger Meza Murillo, Principal Investigator, Multiple Sclerosis Center of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR(AG)05/2023
Record Dates: First submitted 2023-09-05; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, randomized, rater-blinded study (cRHB (N=30) vs RAGT (N=30)).
  For the control group, this protocol includes 24 one-hour sessions of cRHB training during 8 weeks three times per week, under the supervision of a qualified rehab team.
  For the intervention group (RAGT) this protocol includes 24 one-hour sessions of RAGT during 8 weeks three times per week, under the supervision of a qualified rehab team.
  Informed consent will be obtained from patients prior to inclusion in the study, which will be carried out in accordance with the Declaration of Helsinki.
Who Masked: Outcomes Assessor
Masking Description: The eligibility of the subjects from the neurorehabilitation and neurology outpatient clinics of the Multiple Sclerosis Center of Catalonia (Cemcat) will be evaluated.
  And the blinded outcome assessor comes in for just one day to assess each individual, without any information about the therapy that was given to each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Gait Rehabilitation training (tRHB (Active Comparator): Participants randomize to receive a tRHB, will be trained 3 times per week, with an intensity of 40 to 60 minutes, and duration over 8-weeks. Progression will occur by increasing the session intensity weekly.
  A standardized protocol based on the usual clinical practice of physiotherapy in people with multiple sclerosis will be follow, according to patient characteristics, to design the sessions based on the patient objectives to be achieved, choosing the type of specific exercises to be performed based on the patient's condition and with the possibility of adapting them to their evolution during the twenty-four sessions.
  Interventions: Other: tRHB
- Robot Gait training (RAGT): (Experimental): RAGT group, will be trained 3-times per week, with an intensity of 40 to 60 minutes, and duration over 8-weeks. Progression will occur by increasing the session intensity weekly. Training intensity will be monitored and standardized using the Borg Rating of Perceived Exertion scale, and will progress from 'fairly light' to 'somewhat hard'.
  Progression will occur by increasing the number of steps in each session and decrease the level of assistance.
  Participants will be secured with the appropriately sized harness and attached to an overhead body-weight support system. Each session will begin with a 3-5-minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking for up to 30 minutes. During this phase, the force produced by the robot is modulated to support the effort of the patient in producing a typical walking pattern.
  Interventions: Device: Robotic gait training

INTERVENTIONS:
Device: Robotic gait training — RAGT group, will be trained 3-times per week, with an intensity of 40 to 60 minutes, and duration over 8-weeks. Progression will occur by increasing the session intensity weekly. Training intensity will be monitored and standardized using the Borg Rating of Perceived Exertion scale, and will progress from 'fairly light' to 'somewhat hard'.
  Progression will occur by increasing the number of steps in each session and decrease the level of assistance.
  Participants will be secured with the appropriately sized harness and attached to an overhead body-weight support system. Each session will begin with a 3-5-minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking for up to 30 minutes. During this phase, the force produced by the robot is modulated to support the effort of the patient in producing a typical walking pattern.
  Other Names: Robotic; Atalante Gait Training
  Arms: Robot Gait training (RAGT):
Other: tRHB — Participants randomize to receive a tRHB, will be trained 3 times per week, with an intensity of 40 to 60 minutes, and duration over 8-weeks. Progression will occur by increasing the session intensity weekly.
  A standardized protocol based on the usual clinical practice of physiotherapy in people with multiple sclerosis will be follow, according to patient characteristics, to design the sessions based on the patient objectives to be achieved, choosing the type of specific exercises to be performed based on the patient's condition and with the possibility of adapting them to their evolution during the twenty-four sessions.
  Other Names: Physical therapy, gait training
  Arms: Traditional Gait Rehabilitation training (tRHB

SUMMARY:
This trial is a prospective, randomized, rater-blinded study (cRHB (N=30) vs RAGT (N=30)). For the control group, this protocol includes 24 one-hour sessions of cRHB training during 8 weeks three times per week, under the supervision of a qualified rehab team.

For the intervention group (RAGT) this protocol includes 24 one-hour sessions of RAGT during 8 weeks three times per week, under the supervision of a qualified rehab team.

Informed consent will be obtained from patients prior to inclusion in the study, which will be carried out in accordance with the Declaration of Helsinki.

DETAILED DESCRIPTION:
Aims

Primary Aim:

To compare the effect of Robot-Assisted Gait Training (RAGT) using the Atalante self-balance exoskeleton with conventional rehabilitation training (cRHB) for improving Walking speed measured by the Timed 10-meters walk test (10-MWT), considering a clinically relevant change an improvement of 20% of the velocity (m/s) with respect to the baseline assessment.

Secondary Aims:

* To compare the effect of RAGT using the Atalante self-balance exoskeleton with conventional Rehabilitation training (cRHB), for improving static balance, dynamic balance, mobility, and self-perception of gait impairment measured with:

  * Static Balance by the Berg Balance Scale (BBS), considering a clinically relevant change for improvement in balance as measured by BBS was +3 points, meaning that individuals are likely to perceive that as a reproducible and clinically important change in their balance performance.
  * Dynamic balance by the Timed Up and Go test (TUG)
  * Mobility measured by modified Rivermead Mobility Index (mRMI)
  * Self-perception of gait impairment by Multiple Sclerosis Walking Scale-12 (MSWS-12)
  * Instrumented gait analysis by the G-walk device (assessing gait cycle duration, step length, propulsion index, support phase percentage D/I, oscillation phase percentage D/I, double/unique support phase percentage).
* To compare the effect of RAGT using the Atalante self-balance exoskeleton with conventional Rehabilitation training (cRHB) on quality of life, emotional status and fatigue measured at pre and post-intervention with:

  * Multiple Sclerosis Quality of Life-54 (MSQoL 54 Health Survey Spanish version)
  * Hospital Anxiety and Depression Scale (HADs) considering a clinically relevant change of 1.7 points at HADs
  * The Modified fatigue scale (MFIS)
  * The patient' physical effort of each session by means of the scale of perception of the effort R.P.E of Borg at the end of each training.
  * To evaluate the epigenetic blueprint of rehabilitation training by comparing the genome wide chromatin accessibility of peripheral blood mononuclear cells (PBMCs) before and after RAGT or cRHB, by Assay for Transposase-Accessible Chromatin sequencing (ATACseq).
  * To test the hypothesis that genome wide chromatin accessibility compared to clinical measures can be useful for identifying molecular mechanisms underlying rehabilitation therapies.
  * To compare the changes induced by RAGT versus cRHB on the overall chromatin accessibility, and specific genome regions and pathways.
  * Use the biological samples to provide additional functional and mechanistic information about the rehabilitation effects and subject health, disease or state.

Materials And methods

Design:

This trial is a prospective, randomized, rater-blinded study (cRHB (N=30) vs RAGT (N=30)).

For the control group, this protocol includes 24 one-hour sessions of cRHB training during 8 weeks three times per week, under the supervision of a qualified rehab team.

For the intervention group (RAGT) this protocol includes 24 one-hour sessions of RAGT during 8 weeks three times per week, under the supervision of a qualified rehab team.

Additionally, peripheral blood (6ml) will be taken from all subjects at three timepoints: at baseline (T1), after the 8 weeks of rehabilitation treatment (T2) and, if possible, one year after T4. Biological samples will then be given a unique identifier and transferred to researchers for analysis.

Informed consent will be obtained from patients prior to inclusion in the study, which will be carried out in accordance with the Declaration of Helsinki.

Enrollment and Screening Subjects will be evaluated for their eligibility from neurorehabilitation and neurology outpatient clinics at the Multiple Sclerosis Center of Catalonia (Cemcat).

Potential subjects will be referred to the study via Cemcat Physicians. A member of the research team will screen the referral and confirm they meet the necessary inclusion and exclusion criteria. Following confirmation of criteria, potential subjects will be contacted by phone to schedule an initial visit for consent and baseline assessment.

Additionally, peripheral blood (6ml) will also be taken from all subjects at baseline (T1).

Prior to all testing

ELIGIBILITY:
Inclusion Criteria:

* • Male or female, between 18 and 75 years of age.

  * Confirmed diagnosis of MS.
  * EDSS from 6.0 to 7.0.
  * Able to maintain the upright position on a daily basis.
  * Stable course of disease-modifying therapy over the past 6 months.
  * Clinical comorbidity asymptomatic (i.e., no underlying cardiovascular disease)
  * Height: between approximately 1.50 m. and 1.90 m.
  * Willingness to visit the Multiple Sclerosis Center of Catalonia (Cemcat) for testing and training.
  * Gait disorder conditioned by paresis or hemiparesis associated with ataxia or sensory problems.
  * Patient having given written consent.

Atalante is able to accommodate the following limb lengths:

* Thigh: 380-460mm.
* Distance between the ground and the joint space of the knee (to be measured while wearing the shoes they intend to wear with Atalante):

  * 457-607mm for patient with an ankle dorsiflexion ≥ 16°
  * 457-577mm for patient with an ankle dorsiflexion between 13° et 16°
  * 457-567mm for patient with an ankle dorsiflexion between 10° et 13°
  * 457-557mm for patient with an ankle dorsiflexion between 0° and 10°
* Hip with less or equal to 460mm when seated.
* Maximum weight: 90 kg.

Exclusion Criteria:

* • Pregnancy.

  * Starting or switching from fampridine (Fampyra®) in the last 4 weeks.
  * Height and weight outside the secure standard of safe use, described in the safety guides.
  * Contraindications for Atalante training (eg, bone instability, history of osteoporosis or osteoporotic fractures).
  * Subjects under Corticosteroids treatment or relapse.
  * Changes in disease-modifying and symptomatic therapy for MS during the study period.
  * Subjects with psychiatric or cognitive comorbidities that may interfere with the trial.
  * Whose joint centers cannot be aligned Atalante's.
  * Ranges of motion below:

    * Knee: 5° extension, 110° flexion
    * Ankle: 0° dorsiflexion, 9° plantar flexion, 18° inversion and eversion
    * Hip: 115° flexion, 15° extension, 17° abduction, 10° adduction, 10°
    * medial rotation, 20° lateral rotation
  * Severe spasticity (greater than Ashworth 3) or uncontrolled clonus.
  * Severe concurrent medical diseases: infections, circulatory, heart or lung, pressure sores.
  * Active implantable medical device.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Timed 10-meters walk test (10-MWT), | 2 months
  - To compare the effect of RAGT by use of Atalante self-balance exoskeleton with conventional rehabilitation training (cRHB) for improving Walking speed measured by the Timed 10-meters walk test (10-MWT), considering a clinically relevant change an improvement of 20% of the velocity (m/s) with respect to the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Montalban, PHD, Study Director — Multiple Sclerosis Center of Catalonia; Carmen Tur Gomez, PHD, Study Director — Multiple Sclerosis Center of Catalonia
Locations (1):
- Centre d'Esclerosi Mútiple de Catalunya (Cemcat) - Barcelona, Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT06615947/Prot_SAP_000.pdf